CLINICAL TRIAL: NCT05648149
Title: Effect of Preventive Cognitive Training on Cognitive Impairment After Stroke in Acute Stage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023KY757
Record Dates: First submitted 2022-11-23; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-07

CONDITIONS: Stroke, Acute Ischemic; Cognitive Impairment
Keywords: Post-stroke cognitive impairment; stroke; cognitive training; acute stage
MeSH Terms: conditions — Ischemic Stroke; Cognitive Dysfunction; Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hierarchical multi-dimensional cognitive training scheme based on computer (Experimental): Cognitive training was carried out by three trained and certified nurses in accordance with the cognitive training program. Twice a day, 30min each time, for 4 weeks, the difficulty of the training content is divided into 2 levels, the correct rate of more than 80% can enter the next level. During hospitalization, the patients and their families were taught how to use cognitive training programs. After discharge, special personnel were assigned to supervise and urge the patients to carry out cognitive training through the background.
  Interventions: Behavioral: hierarchical multi-dimensional cognitive training scheme based on computer
- routine rehabilitation (No Intervention): Routine treatment, rehabilitation and care

INTERVENTIONS:
Behavioral: hierarchical multi-dimensional cognitive training scheme based on computer — The scheme was constructed five main categories of cognitive function: (1) attention, memory, numeracy, thinking response and perception; (2) There are 10 training items, which are drawing, quick matching, flash memory, number memory, face memory, color tracking, number span, word naming, symbol number form, quick arithmetic; (3) Each training item is divided into basic and advanced training. Only if the basic training reaches more than 80%, can the advanced training be entered; (4) In order to facilitate patient training, all items were embedded in the wechat mini program, and corresponding cognitive training was carried out in the mini program; (5)Small program background can monitor training results.
  Arms: hierarchical multi-dimensional cognitive training scheme based on computer

SUMMARY:
Post-stroke cognitive impairment(PSCI) refers to a clinical syndrome characterized by cognitive impairment that occurs after a stroke event and persists for 6 months. PSCI is divided into post-stroke cognitive impairment non-dementia and post-stroke dementia. About one half of patients develop PSCI within the first year after stroke. Recent large international cohort studies have reported that the incidence of PSCI is 24%-53.4%, among which the incidence of cognitive impairment after stroke without dementia is 14%-29% and the incidence of dementia after stroke is 11%-42%. A study in China shows that the incidence of PSCI is 53.1%. Our previous small sample study also found that the incidence of cognitive impairment in acute phase of ischemic stroke patients was 64.52%. It can be seen that the incidence of PSCI is high, which is an important health problem.

The mortality rate of stroke patients complicated with PSCI is significantly higher than that of patients without cognitive impairment. The 5-year survival rate of patients with post-stroke dementia is only 39%, while the survival rate of stroke patients without dementia of the same age is 75%. In addition, patients with PSCI will lead to long-term disability, a significant decline in self-care ability of daily living, quality of life and mental health status, poor social participation ability, and increased care pressure. If not intervened in time, will bring serious disease and economic burden to the family and society. Therefore, preventing the occurrence and delaying the progression of PSCI is an important task to be solved urgently.

Rehabilitation is an important intervention to delay the progression of PSCI, aiming to promote the remodeling of the central nervous system, and the main method is early and multi-dimensional cognitive function training. Some studies have confirmed that computerization, multi-cognitive domains, and adaptive cognitive training (7 consecutive weeks, 5 days a week, 30 min a day) can significantly improve the global cognitive function of patients with cognitive impairment after subcortical stroke and non-dementia . A recent systematic review showed that cognitive training can improve the cognitive function and daily living ability of patients with mild PSCI. It also has a certain effect on the improvement of patients' overall cognitive function. It can be seen that cognitive training is not effective for all stages of PSCI patients, and the effect of cognitive training is very limited for patients who have developed into a single dimension of severe damage, serious overall cognitive impairment even dementia. This suggests that targeted cognitive intervention for patients at the acute stage of stroke may achieve the purpose of preventing the occurrence and delaying the progression of PSCI.

Therefore, this study innovatively proposed the concept of preventive cognitive training for patients with acute stroke. In the basis of literature research, combined with the views of the cognitive domain experts and Kang Fushi reformed the existing cognitive training plan, build the computer-assisted ladder multidimensional cognitive training scheme, the main dimensions set up on the basis of cognitive training program, according to the degree of cognitive impairment at the same time set the difficulty level of the project, It is convenient for medical staff to select appropriate items and difficulties based on the dimension and degree of cognitive impairment of patients. To evaluate the effect of cognitive training by using cognitive function scale, psycho-psychological scale, self-care ability scale and other tools, and to clarify whether acute preventive cognitive training can improve PSCI, so as to provide a practical basis for the prevention and intervention of PSCI.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed as ischemic stroke by CT or MRI and meeting World Health Organization diagnostic criteria First onset, within 7 days of onset

* There were no contraindications in MRI examination, and the examination was completed with good image quality and complete clinical data
* Between 18 and 64 years old
* Conscious (NIHSS consciousness level 0, 1)
* Informed consent.

Exclusion Criteria:

* Patients with previous cognitive impairment
* Aphasia or severe dysarthria
* Previous cerebral atrophy or white matter lesions
* History of severe cardiopulmonary dysfunction, craniocerebral trauma, etc

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | 0 week
  An assessment tool for rapid screening of cognitive impairment. The total score is 30 points, and the test result shows that the normal value is ≥26 points.
Montreal Cognitive Assessment | 1 week
  An assessment tool for rapid screening of cognitive impairment. The total score is 30 points, and the test result shows that the normal value is ≥26 points.
Montreal Cognitive Assessment | 12 week
  An assessment tool for rapid screening of cognitive impairment. The total score is 30 points, and the test result shows that the normal value is ≥26 points.
Montreal Cognitive Assessment | 24 week
  An assessment tool for rapid screening of cognitive impairment. The total score is 30 points, and the test result shows that the normal value is ≥26 points.
Mini-mental State Examination | 0 week
  n assessment tool for reflect the mental state and the degree of cognitive impairment of the subjects. The total score range of 0-30 points. Scores are closely related to the level of education, and the normal cut-off is defined as: >17 points for illiteracy, >20 points for primary school, and >24 points for junior high school and above.
Mini-mental State Examination | 1 week
  n assessment tool for reflect the mental state and the degree of cognitive impairment of the subjects. The total score range of 0-30 points. Scores are closely related to the level of education, and the normal cut-off is defined as: >17 points for illiteracy, >20 points for primary school, and >24 points for junior high school and above.
Mini-mental State Examination | 12 week
  n assessment tool for reflect the mental state and the degree of cognitive impairment of the subjects. The total score range of 0-30 points. Scores are closely related to the level of education, and the normal cut-off is defined as: >17 points for illiteracy, >20 points for primary school, and >24 points for junior high school and above.
Mini-mental State Examination | 24 week
  n assessment tool for reflect the mental state and the degree of cognitive impairment of the subjects. The total score range of 0-30 points. Scores are closely related to the level of education, and the normal cut-off is defined as: >17 points for illiteracy, >20 points for primary school, and >24 points for junior high school and above.
PSCI Incidence | 12 weeks
  number of PSCI cases/total number of enrolled cases
PSCI Incidence | 24 weeks
  number of PSCI cases/total number of enrolled cases

SECONDARY OUTCOMES:
Hamilton Depression Scale | 0 week
  An assessment tool for assessing depression status. Total score <7: normal; The total score of 7 to 17: depression may be present; The total score of 17 to 24: definitely depression; Total score >24: severe depression.
Hamilton Depression Scale | 1 week
  An assessment tool for assessing depression status. Total score <7: normal; The total score of 7 to 17: depression may be present; The total score of 17 to 24: definitely depression; Total score >24: severe depression.
Hamilton Depression Scale | 12 week
  An assessment tool for assessing depression status. Total score <7: normal; The total score of 7 to 17: depression may be present; The total score of 17 to 24: definitely depression; Total score >24: severe depression.
Hamilton Depression Scale | 24 week
  An assessment tool for assessing depression status. Total score <7: normal; The total score of 7 to 17: depression may be present; The total score of 17 to 24: definitely depression; Total score >24: severe depression.
Hamilton Anxiety Scale | 0 week
  It is mainly used to assess the severity of neurosis and anxiety symptoms in people. A total score of more than 29 may indicate severe anxiety; More than 21 points, there must be significant anxiety; More than 14 points, there is definitely anxiety; More than 7 points, may have anxiety; If the score is less than 7, there are no symptoms of anxiety.
Hamilton Anxiety Scale | 1 week
  It is mainly used to assess the severity of neurosis and anxiety symptoms in people. A total score of more than 29 may indicate severe anxiety; More than 21 points, there must be significant anxiety; More than 14 points, there is definitely anxiety; More than 7 points, may have anxiety; If the score is less than 7, there are no symptoms of anxiety.
Hamilton Anxiety Scale | 12 week
  It is mainly used to assess the severity of neurosis and anxiety symptoms in people. A total score of more than 29 may indicate severe anxiety; More than 21 points, there must be significant anxiety; More than 14 points, there is definitely anxiety; More than 7 points, may have anxiety; If the score is less than 7, there are no symptoms of anxiety.
Hamilton Anxiety Scale | 24 week
  It is mainly used to assess the severity of neurosis and anxiety symptoms in people. A total score of more than 29 may indicate severe anxiety; More than 21 points, there must be significant anxiety; More than 14 points, there is definitely anxiety; More than 7 points, may have anxiety; If the score is less than 7, there are no symptoms of anxiety.
Modified Barthel index | 0 week
  The scale consists of 10 items and 5 different weights of rating scales: unable, attempts but unsafe, moderate help, minimal help, fully independent. There is a score range of 0 to 5 for bathing, grooming; a score range of 0 to 10 for feeding, dressing, bowels, bladder, toilet, stairs; and a score range of 0 to 15 for chair/bed transfers, walking. Higher score represents higher degree of activities daily living independence.
Modified Barthel index | 1 week
  The scale consists of 10 items and 5 different weights of rating scales: unable, attempts but unsafe, moderate help, minimal help, fully independent. There is a score range of 0 to 5 for bathing, grooming; a score range of 0 to 10 for feeding, dressing, bowels, bladder, toilet, stairs; and a score range of 0 to 15 for chair/bed transfers, walking. Higher score represents higher degree of activities daily living independence.
Modified Barthel index | 12 week
  The scale consists of 10 items and 5 different weights of rating scales: unable, attempts but unsafe, moderate help, minimal help, fully independent. There is a score range of 0 to 5 for bathing, grooming; a score range of 0 to 10 for feeding, dressing, bowels, bladder, toilet, stairs; and a score range of 0 to 15 for chair/bed transfers, walking. Higher score represents higher degree of activities daily living independence.
Modified Barthel index | 24 week
  The scale consists of 10 items and 5 different weights of rating scales: unable, attempts but unsafe, moderate help, minimal help, fully independent. There is a score range of 0 to 5 for bathing, grooming; a score range of 0 to 10 for feeding, dressing, bowels, bladder, toilet, stairs; and a score range of 0 to 15 for chair/bed transfers, walking. Higher score represents higher degree of activities daily living independence.
National Institutes of Health Neurological Deficit Score | 0 week
  The scale will assess the degree of the neurological deficit. For all 11 parameters, the top score is 42 points, a score of 0 and 1 is normal, and higher scores mean a worse neurological deficit. We also recorded the neurological deficit result within two days after admission.
National Institutes of Health Neurological Deficit Score | 1 week
  The scale will assess the degree of the neurological deficit. For all 11 parameters, the top score is 42 points, a score of 0 and 1 is normal, and higher scores mean a worse neurological deficit. We also recorded the neurological deficit result within two days after admission.
National Institutes of Health Neurological Deficit Score | 12 week
  The scale will assess the degree of the neurological deficit. For all 11 parameters, the top score is 42 points, a score of 0 and 1 is normal, and higher scores mean a worse neurological deficit. We also recorded the neurological deficit result within two days after admission.
National Institutes of Health Neurological Deficit Score | 24 week
  The scale will assess the degree of the neurological deficit. For all 11 parameters, the top score is 42 points, a score of 0 and 1 is normal, and higher scores mean a worse neurological deficit. We also recorded the neurological deficit result within two days after admission.